CLINICAL TRIAL: NCT04865393
Title: A Phase 1, Open-label Study to Assess the Safety and Pharmacokinetics of SPR206 Following a Single IV Dose of SPR206 in Subjects With Varying Degrees of Renal Function
Brief Title: Phase 1 Study of PK and Safety of SPR206 in Subjects With Various Degrees Of Renal Function
Status: Completed | Phase: Phase 1 | Type: Interventional
Sponsor: Spero Therapeutics (Industry)
Collaborators: United States Department of Defense (U.S. Federal Agency)
Responsible Party: Sponsor
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Other
Other Study IDs: SPR206-103; CDMRP-JW180095-B (Other Grant/Funding Number: United States Department of Defense)
Record Dates: First submitted 2021-04-26; First posted 2021-04-29 (Actual); Last update posted 2024-04-15 (Actual); Status verified 2021-12

CONDITIONS: Renal Impairment
Keywords: End State Renal Disease (ESRD); Renal Insufficiency; Renal Impairment; Renal Disease; Hemodialysis
MeSH Terms: conditions — Renal Insufficiency; Kidney Diseases

STUDY DESIGN:
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (1):
- SPR206 (Experimental): SPR206 100mg single-dose IV infused over 1 hour
  Interventions: Drug: SPR206

INTERVENTIONS:
Drug: SPR206 — SPR206 100 mg single-dose IV infused over 1 hour

SUMMARY:
Evaluation of the pharmacokinetics (PK) of SPR206 in subjects with normal renal function, subjects with various degrees of renal insufficiency, and subjects with end-stage renal disease (ESRD) receiving hemodialysis (HD) therapy.

ELIGIBILITY:
Key Inclusion Criteria:

* BMI ≥ 18.5 and ≤ 39.9 (kg/m2) and weight between 50.0 and 130.0 kg (inclusive)
* Medically healthy without clinically significant abnormalities (Healthy Volunteers) or medically stable without clinically significant acute or chronic illness (Subjects with varying degrees of Renal Disease)
* Normal renal function with eGFR ≥90 mL/min/1.73m2 (Cohort 1), or renal insufficiency with eGFR 60 to <90 mL/min/1.73m2 (Cohort 2), 30 to <60 mL/min/1.73m2 (Cohort 3), or <30 mL/min/1.73m2 (Cohort 4), calculated using Modification of Diet in Renal Disease (MDRD). Subjects with ESRD must be receiving hemodialysis at least 3 times per week for at least 3 months at Screening (Cohort 5 only)
* Non-smoker for at least 1 month prior to screening for the study
* Ability and willingness to abstain from alcohol, caffeine, xanthine-containing beverages or food
* Other inclusion criteria per protocol

Key Exclusion Criteria:

* Any clinically significant medical history or abnormal findings upon physical examination, or clinical laboratory tests, not specifically excluded in other criteria below that, in the opinion of the Investigator, might confound the results of the study or pose an additional risk in administering study drug to the subject
* Electrocardiogram (ECG) with QTcF interval duration equal or greater than 500 msec
* Hemoglobin (HB), hematocrit (HCT), white blood cell count (WBC), or platelet count less than the lower limit of normal range of the reference laboratory (Cohort 1). HB <8.5 gm/dL, WBC ≤3,000 cells/μL or platelet count ≤100,000 cells/μL (Cohorts 2-5)
* Results of biochemistry tests for alanine aminotransferase (ALT), aspartate aminotransferase (AST) and bilirubin greater than 1.5 X the upper limit of normal (ULN) for the reference laboratory
* Recent history (within 6 months) of known or suspected Clostridium difficile infection
* History of chronic liver disease, cirrhosis, or biliary disease
* History of seizure disorder except childhood history of febrile seizures
* Positive urine drug/alcohol testing
* Positive testing for human immunodeficiency virus1/2 (HIV 1/2), hepatitis B surface antigen (HBsAg) or hepatitis C (HCV) antibodies
* History of substance abuse or alcohol abuse
* Known history of clinically significant hypersensitivity reaction or anaphylaxis to any medication
* Other exclusion criteria per protocol

Min Age: 18 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Enrollment: 37 (Actual)
Dates: Start 2021-06-08 (Actual); Primary Completion 2021-12-01 (Actual); Study Completion 2021-12-06 (Actual)

PRIMARY OUTCOMES:
Time to the maximum plasma concentration (Tmax) | 36 hours after start of study drug IV infusion
Maximum plasma concentration (Cmax) | 36 hours after start of study drug IV infusion
Area under the concentration-time curve from time 0 to last measurable timepoint (AUC0-t) | 36 hours after start of study drug IV infusion
Area under the concentration-time curve from time 0 to infinity (AUC0-∞) | 36 hours after start of study drug IV infusion

SECONDARY OUTCOMES:
Area under the concentration-time curve from time 0 to 8 hours (AUC0-8) | 8 hours after start of study drug IV infusion
Terminal Elimination Rate Constant (kel) | 36 hours after start of study drug IV infusion
Terminal half-life (t1/2) | 36 hours after start of study drug IV infusion
Total body clearance (CL) | 36 hours after start of study drug IV infusion
Renal clearance (CLR) | 36 hours after start of study drug IV infusion
Steady-state volume of distribution (Vss) | 36 hours after start of study drug IV infusion
Amount of drug excreted in urine by interval (Aet) for Cohorts 1-4 | 36 hours after start of study drug IV infusion
Cumulative amount of drug excreted in urine at the end of each interval (Aeu) for Cohorts 1-4 | 36 hours after start of study drug IV infusion
Fraction of drug excreted in the urine expressed as a percentage (Ae%) for Cohorts 1-4 | 36 hours after start of study drug IV infusion
Fraction of dose excreted in the urine over a collection interval (Fe) for Cohorts 1-4 | 36 hours after start of study drug IV infusion
Cumulative fraction of dose excreted in the urine over (Feu) for Cohorts 1-4 | 36 hours after start of study drug IV infusion
Extraction ratio (ER) for subjects on dialysis (Cohort 5) | Up to 1 day post dose - between start and end of hemodialysis
Estimated hemodialysis clearance (CLHD) for subjects on dialysis (Cohort 5) | Up to 1 day post dose - between start and end of hemodialysis
Amount of the dose removed by hemodialysis (XHD) for subjects on dialysis (Cohort 5) | Up to 1 day post dose - between start and end of hemodialysis
Incidence of Treatment-Emergent Adverse Events | 14 days post start of last study drug IV infusion
  To assess the incidents of treatment-emergent adverse events following SPR206 intravenous dose administration. AEs will be classified by System Organ Class (SOC) and Preferred Term (PT). Incidence, frequency, severity and duration will be presented.
Incidence of abnormal vital sign assessments - blood pressure | 14 days post study drug IV infusion
  To assess the incidents of abnormal systolic and diastolic blood pressure assessments following SPR206 intravenous dose administration. Values and changes from baseline at each scheduled time-point will be summarized using descriptive statistics (n, mean, SD, median, minimum, and maximum). Significant changes from baseline will be presented.
Incidence of abnormal vital sign assessments - body temperature | 14 days post study drug IV infusion
  To assess the incidents of abnormal body temperature assessments following SPR206 intravenous dose administration. Values and changes from baseline at each scheduled time-point will be summarized using descriptive statistics (n, mean, SD, median, minimum, and maximum). Significant changes from baseline will be presented.
Incidence of abnormal physical exam assessments | 14 days post study drug IV infusion
  To assess the incidents of abnormal body system assessments following SPR206 intravenous dose administration. Changes from baseline in physical examination findings will be classified as Normal, Abnormal NCS, and Abnormal CS. Frequency counts will be presented.
Incidence of abnormal ECG assessments - heart rate | 14 days post study drug IV infusion
  To assess the incidents of abnormal heart rate assessment following SPR206 intravenous dose administration. Cardiac (12-Lead ECG) for heart rate will be classified as normal, abnormality that is NCS, and CS abnormality. Frequency counts by dose group and timepoint of collection will be presented.
Incidence of abnormal ECG assessments - PR, RR, QRS, QT and QTcF interval | 14 days post study drug IV infusion
  To assess the incidents of abnormal PR interval, RR interval, QRS interval, QT interval and QTcF interval assessments following SPR206 intravenous dose administration. Cardiac (12-Lead ECG) results will be classified as normal, abnormality that is NCS, and CS abnormality. Frequency counts by dose group and timepoint of collection will be presented.
Incidence of abnormal safety laboratory assessments | 14 days post study drug IV infusion
  To assess the incidents of abnormal hematology, serum chemistry, coagulation and urinalysis assessments following SPR206 intravenous dose administration. Values and changes from baseline at each scheduled time-point will be summarized using descriptive statistics (n, mean, SD, median, minimum, and maximum). Frequency counts of significant changes from baseline will be presented.

CONTACTS AND LOCATIONS:
Overall Officials: David Melnick, MD, Study Director — Spero Therapeutics Inc
Locations (2):
- New Zealand (2):
  - Medical Facility, Auckland
  - Medical Facility, Christchurch

IPD SHARING:
Plan to Share IPD: No